CLINICAL TRIAL: NCT06278831
Title: Efficacy of Structured SOcial COnsultation and Support in Reducing the FINancial Burden of Radiotherapy
Acronym: SOCOFIN-1
Status: Completed | Type: Observational
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Rami El Shafie, Chief of UMG Radiotherapy, University Medical Center Goettingen
Other Study IDs: 2023-02645
Record Dates: First submitted 2024-01-23; First posted 2024-02-26 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Financial Toxicity
MeSH Terms: conditions — Financial Stress | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Questionnaire — Patients will be approached three times throughout the study at the beforementioned interview dates to fill out a questionnaire. They will be contacted via e-mail, telephone and/or mobile app.

SUMMARY:
Objectives:

* Assess the extent of financial burden of patients undergoing radiotherapy
* Identify clinical and socio-economical factors correlated with the occurrence and extent of financial toxicity
* Design a structured social consultation to reduce financial burden induced by radiotherapy

Inclusion criteria:

1. age ≥ 18 years of age
2. indication for radiation treatment of a malignant disease
3. Karnofsky Performance score (KPS) ≥ 70%
4. Life expectancy ≥ 3 months

Exclusion criteria:

1. Inability to provide informed consent
2. Inability to attend study visits and fulfill data collection requirements
3. Simultaneous participation in other studies which could interfere with this study Primary outcome: Financial burden as expressed by the COST score, measured at baseline and 3 months after completion of radiotherapy

Secondary outcomes:

* Socio-Economic factors at baseline
* Health-related quality of life (EORTC QLQ-C30) at baseline and 3 months
* Depression (PHQ-9) at baseline and 3 months
* Coping mechanisms to address financial burden

Primary Endpoint: Influence of secondary outcomes on changes of the primary outcome (COST-Score) between baseline and 3 months.

Secondary Endpoints:

* Changes in the COST-Score over time
* Changes in PHQ-9 over time
* Changes in EORTC QLQ-C30 over time

This is an exploratory pilot study. To assess the compliance and effectiveness of the used methods all patients willing to participate in the given time period will be enrolled.

To be assessed for eligibility: n = 300 To be allocated/randomised (if applicable) to trial: n = 150 To be analysed: n = 120

DETAILED DESCRIPTION:
The study is designed as a multicenter longitudinal exploratory study of 150 patients. Further details regarding study timetable, inclusion and exclusion criteria and intervention schedule are explained in the destined subsections of this form.

Data is recorded digitally using an electronic case report forms (eCRF). All data is stored pseudonymized in a REDCap® database.

Before enrolment in register, patients will be informed that participation is voluntary and that they may withdraw at any time without having to give reasons and without penalty or loss of benefits to which the subject is otherwise entitled.

In addition, the subject will be given a "Subject Information Sheet", which contains all the important information in writing.

Findings obtained in the course of the cohort study will be stored on electronic media and treated in strict confidence. For the protection of these data, organisational measures have been taken to prevent disclosure to unauthorised third parties.

Background:

Treatment-related financial burden has become increasingly relevant for patients undergoing cancer treatment. Financial burden can encompass several layers, including diminished household income due to the loss of individual working capacity for the duration of treatment and recovery, but also more immediate aspects like the cost of medication, transportation and other out-of-pocket expenses. Those expenses are often either not covered by insurance or need to be paid in advance and later reimbursed, resulting in considerable short-term financial strain. The different aspects of financial burden and their effect on treatment delivery and outcome are summarized under the term "financial toxicity".

Several studies have assessed the effects of financial toxicity on the quality of treatment, as well as on outcomes. They describe the development of coping mechanisms by patients, which could negatively affect treatment adherence and compromise outcomes. Furthermore, deleterious effects on quality of life have been observed as an effect of financial toxicity.

Most of the published literature on financial toxicity has assessed patients treated in the USA, where the amount of treatment-related out-of-pocket expenses can be substantial, depending on the patient's insurance plan. In this model, the lack of insurance coverage for many costly modern treatments can also be a limiting factor to the treatment options a patient can receive, having considerable effect on outcomes in the general population. On the other hand, financial insolvency or debt for the patient and his next of kin can be a result.

Very limited literature is available on the occurrence and effects of financial toxicity in European countries, and Germany in particular, where health insurance is more inclusive and high out-of-pocket expenses for cancer treatment are less likely. Additionally, available literature focuses mainly on patients undergoing drug treatments and little is known about the situation of patients undergoing radiotherapy.

The current study therefore specifically assesses the occurrence and extent of financial toxicity for German cancer patients undergoing radiotherapy treatment. It aims furthermore to identify diagnosis-related and socio-economic risk-factors that can lead to increased financial toxicity, examines coping mechanisms and assesses the effects on health-related quality of life (HR-QoL).

ELIGIBILITY:
Inclusion Criteria:

* cancer diagnosis with indication for radiation
* Karnofsky index minimum 70%
* able to consent
* minimum 18 years old

Exclusion Criteria:

* Inability to provide informed consent
* Inability to attend study visits and fulfill data collection requirements
* Simultaneous participation in other studies which could interfere with this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who are about to receive radiotherapy due to a malignancy are eligible. They must meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2023-07-08 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Financial Toxicity | 4 months
  Measure instrument: Comprehensive Score for financial Toxicity COST score. COST score ranges from 0 (severe) to 44 points (no effect). Primary endpoint: Changes in COST-Score over time. Assessment before radiation therapy, after and 3 months after.

SECONDARY OUTCOMES:
Factors that may influence the occurrence or extent of financial burden | 4 months
  Influence of secondary outcomes on changes of the primary outcome (COST-Score) between baseline and 3 months. Measure instruments:
  - Socio-Economic factors at baseline (highest level of education, salary, type of employment, number of people who contribute to earnings in household, migration background)
Factors that may influence the occurrence or extent of financial burden | 4 months
  Influence of secondary outcomes on changes of the primary outcome (COST-Score) between baseline and 3 months. Measure instruments:
  - Health-related quality of life (EORTC QLQ-C30) at baseline and 3 months: Quality of Life Questionnaire as a Patient-Reported Outcome (PRO) instrument containing 30 questions resulting in multidimensional scores for oncological patients in over 10 subscales
Factors that may influence the occurrence or extent of financial burden | 4 months
  Influence of secondary outcomes on changes of the primary outcome (COST-Score) between baseline and 3 months. Measure instruments:
  - Depression (PHQ-9) at baseline and 3 months: a depressive symptom scale and diagnostic tool to screen adult patients resulting in a score from 0 to 27
Factors that may influence the occurrence or extent of financial burden | 4 months
  Influence of secondary outcomes on changes of the primary outcome (COST-Score) between baseline and 3 months. Measure instruments:
  - Coping mechanisms to address financial burden (economizing, using savings, opening a loan, borrowing money from friends, talking to oncologist about money, not taking medication, non-adherence to therapy, missing appointments, changing therapy regime, applying for financial aid)

CONTACTS AND LOCATIONS:
Overall Officials: Rami El Shafie, Prof. Dr., Principal Investigator — University Medical Center Goettingen; Anna L Kreuser, Study Director — University Medical Center Goettingen
Locations (1):
- University Medical Center Göttingen, Göttingen, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Huntington SF, Weiss BM, Vogl DT, Cohen AD, Garfall AL, Mangan PA, Doshi JA, Stadtmauer EA. Financial toxicity in insured patients with multiple myeloma: a cross-sectional pilot study. Lancet Haematol. 2015 Oct;2(10):e408-16. doi: 10.1016/S2352-3026(15)00151-9. Epub 2015 Sep 17. PMID 26686042
- [Background] Zafar SY, Peppercorn JM, Schrag D, Taylor DH, Goetzinger AM, Zhong X, Abernethy AP. The financial toxicity of cancer treatment: a pilot study assessing out-of-pocket expenses and the insured cancer patient's experience. Oncologist. 2013;18(4):381-90. doi: 10.1634/theoncologist.2012-0279. Epub 2013 Feb 26. PMID 23442307
- [Background] Bestvina CM, Zullig LL, Rushing C, Chino F, Samsa GP, Altomare I, Tulsky J, Ubel P, Schrag D, Nicolla J, Abernethy AP, Peppercorn J, Zafar SY. Patient-oncologist cost communication, financial distress, and medication adherence. J Oncol Pract. 2014 May;10(3):162-7. doi: 10.1200/JOP.2014.001406. PMID 24839274
- [Background] Fenn KM, Evans SB, McCorkle R, DiGiovanna MP, Pusztai L, Sanft T, Hofstatter EW, Killelea BK, Knobf MT, Lannin DR, Abu-Khalaf M, Horowitz NR, Chagpar AB. Impact of financial burden of cancer on survivors' quality of life. J Oncol Pract. 2014 Sep;10(5):332-8. doi: 10.1200/JOP.2013.001322. Epub 2014 May 27. PMID 24865220
- [Background] Ramsey SD, Bansal A, Fedorenko CR, Blough DK, Overstreet KA, Shankaran V, Newcomb P. Financial Insolvency as a Risk Factor for Early Mortality Among Patients With Cancer. J Clin Oncol. 2016 Mar 20;34(9):980-6. doi: 10.1200/JCO.2015.64.6620. Epub 2016 Jan 25. PMID 26811521